CLINICAL TRIAL: NCT02019277
Title: An Open-label, Multicentre, Phase IIIb Study With Intravenous Administration of Pertuzumab, Subcutaneous Trastuzumab, and a Taxane in Patients With HER2-positive Metastatic Breast Cancer
Brief Title: A Study of Pertuzumab and Trastuzumab Subcutaneous (SC) Treatment in Combination With a Taxane in Participants With Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Metastatic Breast Cancer
Acronym: SAPPHIRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28784
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Results first posted 2018-07-23 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; 130-nm albumin-bound paclitaxel; Paclitaxel; pertuzumab; Trastuzumab

ARMS (1):
- Trastuzumab SC, Pertuzumab, and Taxane (Experimental): Participants will receive pertuzumab, trastuzumab and a taxane (docetaxel, paclitaxel or nab-paclitaxel) once every 3 weeks (21-day cycles). Choice of taxane will be at the discretion of the investigator and administered per routine clinical practices and local prescribing instructions.
  Interventions: Drug: Docetaxel; Drug: Nab-paclitaxel; Drug: Paclitaxel; Drug: Pertuzumab; Drug: Trastuzumab

INTERVENTIONS:
Drug: Docetaxel — Dosing regimen to be determined by the investigator, routine clinical practices.
Drug: Nab-paclitaxel — Dosing regimen to be determined by the investigator, routine clinical practices.
Drug: Paclitaxel — Dosing regimen to be determined by the investigator, routine clinical practices.
Drug: Pertuzumab — Pertuzumab will be administered on Day 1 of the first treatment cycle as a loading dose of 840 mg, followed by 420 mg as an IV infusion every 3 weeks.
  Other Names: Perjeta
Drug: Trastuzumab — Trastuzumab will be administered at a fixed dose of 600 mg SC every 3 weeks.
  Other Names: Herceptin

SUMMARY:
This open-label, multicenter, Phase IIIb study will assess the safety, tolerability and efficacy of a combination therapy of intravenous (IV) pertuzumab (Perjeta), trastuzumab (Herceptin) SC, and taxane chemotherapy (docetaxel, paclitaxel or nab-paclitaxel) as first-line therapy in participants with HER2-positive metastatic breast cancer (mBC). All participants will be treated with 3-week cycles of pertuzumab IV (840 milligrams [mg] first dose; subsequent doses of 420 mg) and trastuzumab SC (600 milligrams [mg]). The taxane treatment regimen will be determined by the investigator. Participants will continue therapy until disease progression, unacceptable toxicity, or the participant withdraws consent, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* HER2-positive disease, with an immunohistochemistry score of 3+ or in situ hybridization (ISH)-positive on primary tumor or metastatic site
* Histologically or cytologically confirmed adenocarcinoma of the breast with metastatic disease with at least one measurable lesion and/or non-measurable disease according to RECIST Version 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 for participants who will receive paclitaxel or nab-paclitaxel chemotherapy and ECOG 0-1 for participants who will receive docetaxel chemotherapy
* LVEF of greater than or equal to (>=) 50 percent (%) measured by ECHO or MUGA scan before the first doses of pertuzumab and trastuzumab
* Previous use of either adjuvant or neoadjuvant anti-HER2 therapy is allowed
* Hormonal therapy will be allowed as per institutional guidelines. Hormonal therapy cannot be administered in combination with taxane therapy

Exclusion Criteria:

* Previous systemic non-hormonal anticancer therapy for treatment of mBC
* History of other cancers. Participants with curatively treated carcinoma in situ of the cervix or basal cell carcinoma and participants with other curatively-treated cancers who have been disease-free for at least 5 years are eligible. Participants with previous ductal carcinoma in situ (DCIS) of the breast are also eligible for the study
* Pregnant or breastfeeding women. Positive serum pregnancy test in women of childbearing potential, premenopausal or less than 12 months of amenorrhea post-menopause, within 7 days before the first dose of pertuzumab and trastuzumab
* Current peripheral neuropathy of Grade 3 or greater (National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] Version 4.0)
* Radiographic evidence of central nervous system (CNS) metastases as assessed by computed tomography (CT) or magnetic resonance imaging (MRI), unless they have been treated and have been stable for at least 3 months and do not require ongoing corticosteroid treatment
* Participants with other concurrent serious diseases that may interfere with planned treatment, including severe pulmonary conditions/illness
* Inadequate organ function
* Serious cardiac illness or medical conditions that would preclude the use of trastuzumab
* Participants with severe dyspnea at rest or requiring supplementary oxygen therapy
* Concurrent enrollment in another clinical study using an investigational anti-cancer treatment, within 28 days before the first doses of trastuzumab and pertuzumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-12-05 (Actual); Primary Completion 2016-11-04 (Actual); Study Completion 2016-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (13):
- Australia (13):
  - St George Hospital; Cancer Care Centre, Kogarah, New South Wales
  - Port Macquarie Base Hospital, Port Macquarie, New South Wales
  - Newcastle Mater Misericordiae Hospital; Oncology, Waratah, New South Wales
  - Mater Hospital; Cancer Services, South Brisbane, Queensland
  - Princess Alexandra Hospital Woolloongabba; Clinical Hematology and Medical Oncology, Woolloongabba, Queensland
  - Lyell McEwin Hospital, Adelaide, South Australia
  - Launceston General Hospital, Launceston, Tasmania
  - Bendigo Hospital; Oncology, Bendigo, Victoria
  - Monash Medical Centre; Oncology, Clayton, Victoria
  - Geelong Hospital; Andrew Love Cancer Centre, Geelong, Victoria
  - Royal Melbourne Hospital; Hematology and Medical Oncology, Parkville, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - St John of God Murdoch Hospital; Oncology West, Murdoch, Western Australia

REFERENCES:
- [Derived] Woodward N, De Boer RH, Redfern A, White M, Young J, Truman M, Beith J. Results From the First Multicenter, Open-label, Phase IIIb Study Investigating the Combination of Pertuzumab With Subcutaneous Trastuzumab and a Taxane in Patients With HER2-positive Metastatic Breast Cancer (SAPPHIRE). Clin Breast Cancer. 2019 Jun;19(3):216-224. doi: 10.1016/j.clbc.2019.02.008. Epub 2019 Feb 27. PMID 30922805

RESULTS

PARTICIPANT FLOW:
Groups:
- Trastuzumab, Pertuzumab, and Taxane: Participants received first-line therapy with pertuzumab administered via intravenous (IV) infusion on Day 1 of first treatment cycle (1 cycle = 21 days) at a loading dose of 840 milligrams (mg), followed by 420 mg on Day 1 of each subsequent cycle; trastuzumab administered via subcutaneous (SC) injection at a dose of 600 mg on Day 2 of first treatment cycle, and on Day 1 of each subsequent cycle if both pertuzumab and trastuzumab were well tolerated in Cycle 1; and taxane treatment (docetaxel, paclitaxel, or nabpaclitaxel), administered at the discretion of the investigator, per routine clinical practices and local prescribing instructions. Participants continued study treatment until disease progression (PD), unacceptable toxicity, or withdrawal of consent. Participants with unacceptable toxicity or PD were switched to standard treatment of the investigator's choice. All participants were followed-up until withdrawal of consent, loss to follow-up, death, or study closure.
Period: Overall Study
Arm/Group | Trastuzumab, Pertuzumab, and Taxane
Started | 50
Completed | 38
Not Completed | 12
Not completed — Withdrawal by Subject | 3
Not completed — Death | 7
Not completed — Did no Cooperate | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on the Intent-to-treat (ITT) population, which included all enrolled participants.
Groups:
- Trastuzumab, Pertuzumab, and Taxane: Participants received first-line therapy with pertuzumab administered via IV infusion on Day 1 of first treatment cycle (1 cycle = 21 days) at a loading dose of 840 mg, followed by 420 mg on Day 1 of each subsequent cycle; trastuzumab administered via SC injection at a dose of 600 mg on Day 2 of first treatment cycle, and on Day 1 of each subsequent cycle if both pertuzumab and trastuzumab were well tolerated in Cycle 1; and taxane treatment (docetaxel, paclitaxel, or nabpaclitaxel), administered at the discretion of the investigator, per routine clinical practices and local prescribing instructions. Participants continued study treatment until PD, unacceptable toxicity, or withdrawal of consent. Participants with unacceptable toxicity or PD were switched to standard treatment of the investigator's choice. All participants were followed-up until withdrawal of consent, loss to follow-up, death, or study closure.
Arm/Group | Trastuzumab, Pertuzumab, and Taxane
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious AEs
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Percentage of participants with AEs and SAEs was reported. AEs included both SAEs and non-SAEs. The 95% confidence interval (CI) was computed using Clopper-Pearson method.
Time Frame: Baseline up to 28 days after last study drug administration (up to 36 months)
Population: Analysis was performed on the Safety population, which included all enrolled participants who received at least one dose of pertuzumab IV or trastuzumab SC.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab, Pertuzumab, and Taxane
Number analyzed (Participants) | 50
percentage of participants
  AEs | 100.0 [92.9 to 100.0]
  SAEs | 54.0 [39.3 to 68.2]

2. Secondary Outcome: Percentage of Participants With Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: BOR was defined as a confirmed CR or PR. All measurable lesions up to a maximum of 2 lesions per organ and 5 in total were identified as target lesions (TLs) and recorded at baseline. A sum of the diameters (longest for non-nodal lesions, short axis [SA] for nodal lesions) for all TLs was calculated as baseline sum of diameters (SD). All other lesions (or sites of disease) were identified as non-TLs and were recorded at baseline. CR was defined as the disappearance of all TLs and SA reduction to less than (<) 10 millimeter (mm) for nodal TLs/ non-TLs. PR was defined as greater than or equal to (>/=) 30% decrease in SD of TLs, taking as reference the baseline SD. Confirmation of response at a consecutive tumor assessment at least 4 weeks apart was required. The 95% CI was computed using Clopper-Pearson method.
Time Frame: Baseline up to withdrawal of consent, loss to follow-up, disease progression, death, or study end (up to approximately 36 months)
Population: Analysis was performed on ITT population. Only participants with measurable disease at baseline were included in the analysis. Participants without a post-baseline tumor assessment were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab, Pertuzumab, and Taxane
Number analyzed (Participants) | 45
percentage of participants | 73.3 [58.1 to 85.4]

3. Secondary Outcome: Percentage of Participants With PD (Assessed According to RECIST Version 1.1) or Death Due to Any Cause
Description: For TLs, PD was defined as >/=20% relative increase and >/=5 mm of absolute increase in the SD, taking as reference the smallest SD recorded since treatment started or the appearance of 1 or more new lesions. For non-TLs, PD was defined as appearance of 1 or more new lesions and/or unequivocal progression of existing non-TLs.
Time Frame: as for outcome 2
Population: Analysis was performed on the ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab, Pertuzumab, and Taxane
Number analyzed (Participants) | 50
percentage of participants | 60.0 [58.1 to 85.4]

4. Secondary Outcome: Progression-free Survival (PFS) Assessed According to RECIST Version 1.1
Description: PFS was defined as the time from start of treatment until first documented PD or death from any cause, whichever occurred first. Participants without PD, death, or who were lost to follow-up at the time of analysis were censored at the date of the last tumor assessment when non-progression was documented or at the last date of follow-up, whichever was last. Participants without tumor assessment data after the baseline were censored at baseline unless death occurred before first scheduled tumor assessment. PD was defined as >/=20% relative increase and >/=5 mm of absolute increase in the SD of TLs, taking as reference the smallest SD recorded since treatment started, and/or unequivocal progression of existing non-TLs, or appearance of 1 or more new lesions. Median PFS was estimated using Kaplan-Meier method. The 95% CI was computed using Brookmeyer and Crowley method.
Time Frame: as for outcome 2
Population: Analysis was performed on the ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab, Pertuzumab, and Taxane
Number analyzed (Participants) | 50
months | 17.02 [12.48 to 31.18]

5. Secondary Outcome: Percentage of Participants Who Died Due to Any Cause
Description: Percentage of participants who died due to any cause during the study was reported.
Time Frame: as for outcome 2
Population: Analysis was performed on the ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab, Pertuzumab, and Taxane
Number analyzed (Participants) | 50
percentage of participants | 18.0 [58.1 to 85.4]

6. Secondary Outcome: Overall Survival (OS)
Description: The OS was defined as the time from the start of treatment until death from any cause. Participants alive at the time of analysis and participants who were lost to follow-up were censored at their last clinical assessment date. Median OS was estimated using Kaplan-Meier method. The 95% CI was computed using Brookmeyer and Crowley method.
Time Frame: as for outcome 2
Population: Analysis was performed on the ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab, Pertuzumab, and Taxane
Number analyzed (Participants) | 50
months | NA [31.28 to NA] — Median and Upper Limit for 95% CI could not be estimated due to high number of censored participants.

7. Secondary Outcome: Event-free Survival (EFS) Assessed According to RECIST Version 1.1
Description: EFS was defined as the time from the start of treatment until the first documented initiation of non-protocol-specified treatment for metastatic breast cancer, PD, or death from any cause, whichever occurred first. Participants without treatment change, PD, death, or who were lost to follow-up at the time of analysis were censored at the date of the last tumor assessment when non-progression was documented or at the last date of follow-up, whichever was last. Participants without tumor assessment after baseline were censored at baseline unless death occurred before first scheduled tumor assessment. PD was defined as >/=20% relative increase and >/=5 mm of absolute increase in the SD of TLs, taking as reference the smallest SD recorded since treatment started, and/or unequivocal progression of existing non-TLs, or appearance of 1 or more new lesions. Median EFS was estimated using Kaplan-Meier method. The 95% CI was computed using Brookmeyer and Crowley method.
Time Frame: as for outcome 2
Population: Analysis was performed on the ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab, Pertuzumab, and Taxane
Number analyzed (Participants) | 50
months | 17.02 [12.48 to 31.18]

8. Secondary Outcome: Percentage of Participants Who Died During Receiving Second-Line of Treatment
Description: Percentage of participants who died from any cause during second-line of treatment was reported.
Time Frame: From start of second-line of treatment (any time from baseline up to 35 months) up to death due to any cause or study end (up to approximately 36 months)
Population: Analysis was performed on the ITT population participants who started second-line of treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab, Pertuzumab, and Taxane
Number analyzed (Participants) | 30
percentage of participants | 30.0 [58.1 to 85.4]

9. Secondary Outcome: OS During Second-Line of Treatment
Description: The OS during second-line therapy was defined as the time from the start of second-line therapy (failure of first-line therapy) until death from any cause. Participants alive at the time of analysis and participants who were lost to follow-up were censored at their last clinical assessment date. Median OS during second-line therapy was estimated using Kaplan-Meier method. The 95% CI was computed using Brookmeyer and Crowley method.
Time Frame: as for outcome 8
Population: Analysis was performed on the ITT population participants who started second-line of treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab, Pertuzumab, and Taxane
Number analyzed (Participants) | 30
months | 21.29 [14.85 to 29.04]

10. Secondary Outcome: Number of Participants Receiving Second-Line Treatment by Treatment Type
Description: Second-line anti-cancer treatment was initiated after disease progression on first-line therapy. Number of participants who started second-line of treatment by treatment type was reported. Participants who received combination treatment were counted for each treatment type.
Time Frame: Baseline up to approximately 35 months
Population: Analysis was performed on the ITT population participants who started second-line of treatment.
Measure: Number; unit: participants
Arm/Group | Trastuzumab, Pertuzumab, and Taxane
Number analyzed (Participants) | 30
participants
  Capecitabine | 8 [58.1 to 85.4]
  Cyclophosphamide | 2
  Denosumab | 2
  Doxorubicin | 1
  Epirubicin | 1
  Eribulin | 1
  Fluorouracil | 1
  Lapatinib | 4
  Nanoparticle Paclitaxel | 1
  Paclitaxel | 4
  Pertuzumab | 5
  Trastuzumab | 13
  Trastuzumab Emtansine | 10
  Vinorelbine | 1

11. Primary Outcome: Percentage of Participants With AEs by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.0 Intensity Grades
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Intensity of AEs were graded according to NCI CTCAE version 4.0 on a 5-point scale: Grade 1=Mild, intervention not indicated; Grade 2=Moderate, local or noninvasive intervention indicated; Grade 3=Severe or medically significant but not immediately life-threatening; Grade 4= Life-threatening consequences, urgent intervention indicated; and Grade 5=Death related to AE. Percentage of participants with AEs by maximum severity grades was reported.
Time Frame: Baseline up to 28 days after last study drug administration (up to 36 months)
Population: Analysis was performed on the Safety population.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab, Pertuzumab, and Taxane
Number analyzed (Participants) | 50
percentage of participants
  Grade 1 | 4.0 [92.9 to 100.0]
  Grade 2 | 32.0 [39.3 to 68.2]
  Grade 3 | 50.0
  Grade 4 | 12.0
  Grade 5 | 2.0

12. Primary Outcome: Percentage of Participants With AEs Leading to Premature Discontinuation of Investigational Medicinal Products (IMPs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Percentage of participants with AEs leading to premature discontinuation of IMPs (pertuzumab and trastuzumab) was reported. AEs included both SAEs and non-SAEs. The 95% CI was computed using Clopper-Pearson method.
Time Frame: Baseline up to 28 days after last study drug administration (up to 36 months)
Population: Analysis was performed on the Safety population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab, Pertuzumab, and Taxane
Number analyzed (Participants) | 50
percentage of participants | 12.0 [4.5 to 24.3]

13. Primary Outcome: Percentage of Participants With AEs of Suspected Cardiac Origin, by New York Heart Association Classification (NYHA)
Description: NYHA functional classification includes: Class I (no limitation in physical activity; ordinary physical activity does not cause fatigue, breathlessness or palpitation), Class II (slight limitation of physical activity; ordinary physical activity results in fatigue, palpitation, breathlessness or angina pectoris), Class III (marked limitation of physical activity; less than ordinary activity will lead to symptomatically 'moderate' heart failure) and Class IV (inability to carry out any physical activity without discomfort; symptoms of congestive cardiac failure are present even at rest). Percentage of participants with AEs suspected to be of cardiac origin by maximum NYHA classification was reported.
Time Frame: Baseline up to 28 days after last study drug administration (up to 36 months)
Population: Analysis was performed on the Safety population.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab, Pertuzumab, and Taxane
Number analyzed (Participants) | 50
percentage of participants
  Class I | 6.0 [4.5 to 24.3]
  Class II | 4.0
  Class III | 2.0
  Class IV | 0.0

14. Primary Outcome: Percentage of Participants With Left Ventricular Ejection Fraction (LVEF) Below 50%
Description: LVEF was assessed using echocardiography (ECHO) or multiple-gated acquisition (MUGA) scans. Percentage of participants with LVEF below 50% at any time during the study was reported.
Time Frame: Baseline up to 28 days after last study drug administration (up to 36 months)
Population: Analysis was performed on the Safety population.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab, Pertuzumab, and Taxane
Number analyzed (Participants) | 50
percentage of participants | 8.0

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last study drug administration (up to 36 months)
Arm/Group | Trastuzumab, Pertuzumab, and Taxane
Serious Adverse Events (participants affected / at risk) | 27/50
Other Adverse Events (participants affected / at risk) | 49/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab, Pertuzumab, and Taxane (N=50)
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Anaemia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 7
Mucosal inflammation (General disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Cellulitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Device related infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Syncope (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab, Pertuzumab, and Taxane (N=50)
Anaemia (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 8
Tachycardia (Cardiac disorders) | 3
Dry eye (Eye disorders) | 6
Lacrimation increased (Eye disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 9
Diarrhoea (Gastrointestinal disorders) | 35
Dry mouth (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 12
Nausea (Gastrointestinal disorders) | 23
Stomatitis (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 17
Chest discomfort (General disorders) | 3
Chest pain (General disorders) | 3
Chills (General disorders) | 4
Fatigue (General disorders) | 34
Injection site reaction (General disorders) | 3
Mucosal inflammation (General disorders) | 5
Oedema peripheral (General disorders) | 4
Pain (General disorders) | 3
Conjunctivitis (Infections and infestations) | 3
Nail infection (Infections and infestations) | 3
Oral candidiasis (Infections and infestations) | 4
Paronychia (Infections and infestations) | 7
Rash pustular (Infections and infestations) | 4
Sinusitis (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 19
Urinary tract infection (Infections and infestations) | 10
Weight decreased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 6
Hypocalcaemia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 12
Back pain (Musculoskeletal and connective tissue disorders) | 10
Bone pain (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 14
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 18
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11
Dizziness (Nervous system disorders) | 9
Dysgeusia (Nervous system disorders) | 7
Headache (Nervous system disorders) | 17
Lethargy (Nervous system disorders) | 5
Neuropathy peripheral (Nervous system disorders) | 28
Peripheral sensory neuropathy (Nervous system disorders) | 5
Anxiety (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4
Acne (Skin and subcutaneous tissue disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 27
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 8
Erythema (Skin and subcutaneous tissue disorders) | 4
Nail disorder (Skin and subcutaneous tissue disorders) | 12
Pruritus (Skin and subcutaneous tissue disorders) | 7
Rash (Skin and subcutaneous tissue disorders) | 26
Skin lesion (Skin and subcutaneous tissue disorders) | 3
Tooth extraction (Surgical and medical procedures) | 3
Hot flush (Vascular disorders) | 7
Hypertension (Vascular disorders) | 6
Lymphoedema (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.